CLINICAL TRIAL: NCT06045273
Title: The Elders' Resilience Curriculum: Toward Building Empirical Evidence Around a Culturally-Grounded, Strengths-Based Intervention
Brief Title: The Elders' Resilience Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00018615; K01MH122702 (NIH)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Suicidal Ideation
Keywords: American Indian; Alaska Native; Suicide prevention
MeSH Terms: conditions — Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elders' Resilience Curriculum Recipients (Experimental): Youth aged 9-14 who receive the Elders' Resilience Curriculum
  Interventions: Behavioral: Elders' Resilience Curriculum

INTERVENTIONS:
Behavioral: Elders' Resilience Curriculum — The Elders' Resilience Curriculum (ERC) is a culturally grounded, school-based program taught by White Mountain Apache Tribe (WMAT) Elders to youth. It is designed to prevent suicide ideation and behaviors for American Indian youth
  Other Names: ERC

SUMMARY:
The overall goal of this research is to better understand if and how the Elders' Resilience Curriculum (ERC), a culturally grounded, school-based upstream suicide prevention program taught by White Mountain Apache Tribe (WMAT) Elders to youth, promotes connectedness, cultural strengths, and reasons for living among American Indian youth.

DETAILED DESCRIPTION:
The overall goal of this research is to better understand if and how the Elders' Resilience Curriculum (ERC), a culturally grounded, school-based upstream suicide prevention program taught by White Mountain Apache Tribe (WMAT) Elders to youth, promotes connectedness, cultural strengths, and reasons for living among American Indian youth. Prior to this trial, the investigators collaborated with WMAT research partners to gather qualitative data to identify key protective factors and core components of the ERC. After identifying key protective factors and core components of the ERC, the investigators developed a culturally adapted assessment battery and theoretical model to assess the ERC. This study works with White Mountain Apache tribal community partners to collaboratively pilot test a rigorous evaluation of the ERC.

ELIGIBILITY:
Inclusion Criteria:

* Ages 9-14 years
* Enrolled in a school where the Elders' Resilience Curriculum is delivered
* Participating in the Elders' Resilience Curriculum Program

Exclusion Criteria:

* Parent/Guardian objection to youth participation

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria O'Keefe, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- CIH Whiteriver Office, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elders' Resilience Curriculum Recipients
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elders' Resilience Curriculum Recipients
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (1.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 72
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Reasons for Life as Assessed by the Reasons for Life Scale
Description: 11 self-report items from the Reasons for Life scale, measures beliefs and experiences that make youth feel like life is enjoyable, worthwhile, and meaningful. Responses range from 1 (not at all) to 3 (a lot) with higher scores indicating more reasons for life. Total scores range from 11-33 with higher scores indicating more reasons for life. Change was calculated from the difference between endline and baseline responses.
Time Frame: Baseline, 26 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Elders' Resilience Curriculum Recipients
Number analyzed (Participants) | 72
score on a scale | 2.36 (0.0351)
Statistical Analysis 1: Comparison: Elders' Resilience Curriculum Recipients; Test type: Superiority; p = 0.0006, Satterthwaite approximations; Also used a mixed models analysis; Slope = 0.224, Standard Error of Mean 0.064

2. Primary Outcome: Change in Cultural Connectedness as Assessed by the Cultural Connectedness Scale - Short Form
Description: The Cultural Connectedness Scale-short version is a 9-item self-report measure that assesses connection to cultural identity, traditions, and spirituality among First Nations youth. Responses vary - five questions are yes/no, three questions range from 0 (disagree) to 1 (agree) and the last question ask about frequency, ranging from 0 (never) to 4 (every day). Higher agreement (i.e., "yes" or "agree" responses) indicate greater levels of cultural connectedness. Total scores range from 0-12 with higher scores indicating greater levels of cultural connectedness. Change was calculated from the difference between endline and baseline responses.
Time Frame: Baseline, 26 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Elders' Resilience Curriculum Recipients
Number analyzed (Participants) | 72
score on a scale | 0.756 (0.0217)
Statistical Analysis 1: Comparison: Elders' Resilience Curriculum Recipients; Test type: Superiority; p = 0.0504, Satterthwaite approximations; Also used a mixed models analysis; Slope = 0.084, Standard Error of Mean 0.043

3. Secondary Outcome: Change in Awareness of Connectedness as Assessed by the Awareness of Connectedness Scale
Description: The Awareness of Connectedness Scale is a 12-item self-report measure that evaluates awareness of connection with self, family, community, and the natural environment. Responses range from 0 (not at all) to 2 (a lot) with higher scores representing greater levels of awareness of connectedness. Total scores range from 0-24 with higher scores representing greater levels of awareness of connectedness. Change was calculated from the difference between endline and baseline responses.
Time Frame: Baseline, 26 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Elders' Resilience Curriculum Recipients
Number analyzed (Participants) | 72
score on a scale | 1.04 (0.0394)
Statistical Analysis 1: Comparison: Elders' Resilience Curriculum Recipients; Test type: Superiority; p = 0.00134, Satterthwaite approximations; Also used a mixed models analysis; Slope = 0.131, Standard Error of Mean 0.04

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Elders' Resilience Curriculum Recipients
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT06045273/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT06045273/ICF_001.pdf